CLINICAL TRIAL: NCT04048759
Title: The Promotion of Physical Activity for the Prevention of Alzheimer's Disease in Adults With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00143836; R01AG063909 (NIH)
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Down Syndrome; Alzheimer Disease
Keywords: Physical Activity; Exercise
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remote Low (Other)
  Interventions: Behavioral: Remote Low
- Remote High (Other)
  Interventions: Behavioral: Remote High
- Personal Coach (Other)
  Interventions: Behavioral: Personal Coach

INTERVENTIONS:
Behavioral: Remote Low — Participants will attend 40 min remotely delivered group MVPA sessions once a week, receive a step counter, access to resources for increasing MVPA, and one 20-min remotely delivered individual support/education session/wk.
  Arms: Remote Low
Behavioral: Remote High — Participants will attend 40 min remotely delivered group MVPA sessions 3x a week, receive a step counter, access to resources for increasing MVPA, and one 20-min remotely delivered individual support/education session/wk.
  Arms: Remote High
Behavioral: Personal Coach — Participants will receive a step counter, access to resources for increasing MVPA, and monthly remote individual support/education.
  Arms: Personal Coach

SUMMARY:
The objectives of this study are to determine the feasibility and potential efficacy of remotely delivered group exercise sessions to increase daily moderate to vigorous physical activity in adults with Down syndrome, relative to a usual care control. Participants will be randomized to attend 40 min remotely delivered group moderate to vigorous physical activity (MVPA) sessions at low frequency (1 session/wk.,RL), high frequency (3 sessions/wk., RH), or usual care control usual care control (UC). In addition to the group MVPA sessions, participants in both the RL and RH groups will also receive a step counter, access to resources for increasing MVPA, and one 20-min remotely delivered individual support/education session/wk. Content for both the RL and RH arms will be identical with the exception of group session frequency (1 vs. 3/wk.). Participants in the UC arm will receive a step counter, access to resources for increasing MVPA, and monthly remote individual support/education).The primary aim is to Assess daily MVPA (min) in the RL, RH, and UC arms at baseline, 3, 6, 9, and 12 mos., and obtain effect sizes for change in MVPA over 12-mos.Secondary Aim 1 is to assess the impact of MVPA on cardiovascular fitness, quality of life, cognitive function, and brain parameters related to Alzheimer's Disease (whole and regional brain volume, functional connectivity, and cerebral blood flow) at baseline, 6, and 12 mos. Secondary Aim 2 will determine the feasibility (retention, session attendance, use of recorded sessions (RH/RL only) of RL, RH, and UC interventions.

DETAILED DESCRIPTION:
This research study will compare 3 strategies for the delivery of an intervention to increase moderate to vigorous physical activity (MVPA) in community dwelling adults with Down Syndrome; remotely delivered group MVPA sessions at low (1 session/wk.,RL), high frequency (3 sessions/wk., RH), or usual care control (UC). Adults (age ≥ 18 yrs.) with Down Syndrome will be randomized (2:2:1) to one of the 3 intervention arms for an 12-mo. trial. Cohorts of ~20 adults with Down Syndrome will be recruited and computer randomized. Participants will be stratified by sex and sequentially randomized by the study statistician. Participants in all arms will be provided with an iPad for intervention delivery, Fitbit for self-monitoring MPA, and will be asked to complete 150 min of MPA/wk. Participants in the RL and RH arms will be asked to complete 40 minutes MVPA sessions delivered via Zoom software on an iPad, RL will be provided 1 session/wk, and RH will be provided 3 sessions/wk. Participants in both the RL and RH groups will also receive one 20-min remotely delivered individual support/education session/wk. with a heath coach to discuss progress and provide support. The UC intervention will follow the traditional approach to promote increased MVPA. Participants will receive an iPad tablet loaded with information regarding increasing MVPA and will also receive resistance bands and a Fitbit for self-monitoring MVPA. Monthly 20-min. education/support sessions, identical to the education/support sessions provided in the RL and RH arms, will be delivered to participants and their caregivers remotely on the iPad using FaceTime. All outcomes will be collected by trained research assistants who are blinded to the study condition. The primary outcome, daily MVPA (min) in the RL, RH, and UC arms will be assessed at baseline, 3, 6, 9, and 12 mos. using an accelerometer. All secondary outcomes will be assessed at baselines, 6, and 12 months. Secondary outcomes are to assess the impact of MVPA across the RL, RH, and UC arms on cardiovascular fitness, quality of life, cognitive function and brain parameters related to Alzheimer's Disease (whole and regional brain volume, functional connectivity, cerebral blood flow). Additionally the researchers will determine the feasibility (retention, session attendance, use of recorded sessions (RH/RL only) and safety of RL, RH, and UC arms.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and over.
* Diagnosis of DS as determined by a Community Service Provider operating in our recruitment area under the auspices of a Community Developmental Disability Organization (CDDO).
* Sufficient functional ability to understand directions, communicate preferences, wants and needs through spoken language.
* Living at home with a parent/guardian or in a supported living environment with a caregiver who agrees to serve as a study partner.
* No plans to relocate outside the study area over the next 12 mos.
* Internet access in the home.

Exclusion Criteria:

* Diagnosis of dementia as determine by the Cambridge Examination for Mental Disorders of Older People with Down Syndrome and others with intellectual disabilities.
* Unable to participate in MVPA.
* Pregnancy during the previous 6 mos., currently lactating or planned pregnancy in the following 12 mos.
* Serious medical risk, e.g., cancer, recent heart attack, stroke, angioplasty as determined by the PCP.
* Unwilling to be randomized.
* Participation in a regular exercise program, i.e. greater than or equal to 20 min/d greater than or equal to 3 d/wk.
* Contraindications for MRI, including metal implants or devices incompatible with MRI such as pacemakers, claustrophobia, and inability to lay in a supine position.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Ptomey, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ptomey LT, Helsel BC, Washburn RA, Montgomery RN, Krebill R, Danon JC, Sherman JR, Forsha D, Bodde A, Szabo-Reed AN, Gorczyca AM, Donnelly JE. The promotion of physical activity for use in Alzheimer's disease prevention trials in adults with Down syndrome: Results from a 12-month randomized trial. Alzheimers Dement (N Y). 2025 Jun 12;11(2):e70115. doi: 10.1002/trc2.70115. eCollection 2025 Apr-Jun. PMID 40520478
- [Derived] Frank L, Helsel B, Dodd D, Bodde AE, Danon JC, Sherman JR, Forsha DE, Szabo-Reed A, Washburn RA, Donnelly JE, Ptomey LT. The association between cardiovascular health and cognition in adults with Down syndrome. J Neurodev Disord. 2023 Dec 6;15(1):43. doi: 10.1186/s11689-023-09510-z. PMID 38057709
- [Derived] Dodd D, Helsel B, Bodde AE, Danon JC, Sherman JR, Donnelly JE, Washburn RA, Ptomey LT. The association of increased body mass index on cardiorespiratory fitness, physical activity, and cognition in adults with down syndrome. Disabil Health J. 2023 Oct;16(4):101497. doi: 10.1016/j.dhjo.2023.101497. Epub 2023 Jun 16. PMID 37407386
- [Derived] Ptomey LT, Szabo-Reed AN, Martin LE, Mayo MS, Washburn RA, Gorczyca AM, Lepping RJ, Lee P, Forsha DE, Sherman JR, Danon JC, Donnelly JE. The promotion of physical activity for the prevention of Alzheimer's disease in adults with Down Syndrome: Rationale and design for a 12 Month randomized trial. Contemp Clin Trials Commun. 2020 Jun 30;19:100607. doi: 10.1016/j.conctc.2020.100607. eCollection 2020 Sep. PMID 32642594

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remote High | Remote Low | Personal Coach
Started | 34 | 32 | 15
6 Month Assessment | 34 | 32 | 15
12 Month Assessment | 34 | 32 | 15
Completed | 34 | 32 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remote High | Remote Low | Personal Coach | Total
Number analyzed (Participants) | 34 | 32 | 15 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (8.5) | 27.8 (10.4) | 26.6 (6.6) | 26.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 7 | 45
  Male | 15 | 13 | 8 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 1 | 7
  Not Hispanic or Latino | 31 | 29 | 14 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 2 | 3 | 0 | 5
  White | 32 | 21 | 15 | 68
  More than one race | 0 | 4 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 32 | 15 | 81

OUTCOME MEASURES:

1. Primary Outcome: Minutes of Moderate to Vigorous Physical Activity (MVPA) Per Day
Description: MVPA was assessed using an ActiGraph tri-axial accelerometer.
Time Frame: Baseline to 12 months
Population: Only participants who had valid accelerometer wear time (8 hrs a day for at least 3 weekdays/1weekend day) are included at each timepoint.
Measure: Mean (Standard Deviation); unit: min of MVPA/day
Arm/Group | Remote High | Remote Low | Personal Coach
Number analyzed (Participants) | 34 | 32 | 15
min of MVPA/day
  Absolute MVPA at Baseline: number analyzed (Participants) | 27 | 28 | 12
  Absolute MVPA at Baseline | 13.8 (13.9) | 17.9 (29.6) | 15.6 (15.8)
  Absolute MVPA at 3 months: number analyzed (Participants) | 31 | 26 | 10
  Absolute MVPA at 3 months | 21.8 (19.3) | 13.8 (12.6) | 19.9 (18.3)
  Absolute MVPA at 6 months: number analyzed (Participants) | 30 | 26 | 11
  Absolute MVPA at 6 months | 26.1 (24.4) | 15.9 (15.7) | 20.0 (18.6)
  Absolute MVPA at 9 months: number analyzed (Participants) | 32 | 29 | 12
  Absolute MVPA at 9 months | 23.9 (21.4) | 19.5 (24.9) | 17.9 (17.0)
  Absolute MVPA at 12 months: number analyzed (Participants) | 30 | 29 | 12
  Absolute MVPA at 12 months | 24.4 (23.5) | 14.7 (16.7) | 17.0 (13.9)

2. Secondary Outcome: Cognitive Function
Description: Working memory, processing speed, multitasking, and episodic memory will be assessed at baseline, 6 and, and 12 months, using tests selected from the widely used Cambridge Neuropsychological Test Automated Battery (CANTAB, Cambridge Cognition, LTD, Cambridge, UK) for Down syndrome. The CANTAB for Down syndrome uses a battery of tests including multitasking, episodic memory, executive function and processing speed.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Cardiovascular Fitness
Description: Maximal treadmill tests (modified Balke protocol) will be completed at baseline, 6, and 12 months
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Change in Quality of Life
Description: Quality of life will be assessed at baseline, 6, and 12 months with the Personal Well-Being Index Intellectual Disability, which contains 7 items, each corresponding to a quality of life domain: standard of living, health, life achievement, personal relationships, personal safety, community connectedness, and future security. Participants answer questions on a 0-4 scale, with 0 being least happy and 4 being most happy.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Brain Volume
Description: Brain volume will be measured using structural MRI at baseline, 6, and 12 months
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Functional Connectivity
Description: Functional connectivity will be measured using resting state MRI (rsMRI) at baseline, 6, and 12 months.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

7. Secondary Outcome: Cerebral Blood Flow
Description: Functional connectivity will be measured using arterial spin labeling at baseline, 6, and 12 months
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

8. Secondary Outcome: Retention
Description: Retention will be measured by the percentage of participants who complete the 12 month intervention, defined as completing the 12 month outcome assessments.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

9. Secondary Outcome: Session Attendance
Description: Session attendance for both group MVPA and education/support sessions from baseline to 12 months will be obtained from records maintained by the health educator, and expressed as the percent of possible sessions. Attendance at group MVPA sessions will be defined as being logged in to the video conference and remaining on the screen for the entire 30-min session. Attendance at individual support/education sessions, for the both exercise and UC conditions, will be defined as answering the FaceTime call, and being present on screen for the entire session.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

10. Secondary Outcome: Use of Recorded Exercise Sessions
Description: Use of recorded exercise sessions will be tracked using Dropbox which provides information on how many times each user watched a video.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

11. Secondary Outcome: Reported Serious Adverse Event
Description: Safety will be measured by number of participants reporting a serious adverse event, i.e., any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or results in persistent or significant disability/incapacity.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Weight
Description: Weight will be measured in light clothing on a calibrated scale (Model #PS6600, Belfour, Saukville, WI) to the nearest 0.1 kg.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Height
Description: Standing height will be measured with a portable stadiometer (Model #IP0955, Invicta Plastics Limited, Leicester, UK).
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Waist Circumference
Description: Waist circumference will be assessed using a waist tape measure.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Energy Expenditure of Exercise Sessions
Description: The energy expenditure of sessions will be collected by a portable metabolic system at random timepoints across the 12 month study.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Functional Lower Extremity Strength
Description: Functional lower extremity strength will be assessed using the Five Times Sit to Stand
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Functional Mobility
Description: Functional mobility will be assessed using the Timed Up and Go.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Upper Body Strength
Description: Upper body strength will be assessed using hand grip dynamometer
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Activities of Daily Living
Description: Activities of daily living will be assessed using the Waisman Activities of Daily Living scale. This scale contains 17 questions, each item is rated as 0="does not do", 1="does with help", or 2="does independently / on own. A higher score indicates greater independence.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Caregiver Burden
Description: Caregiver burden will be assess using The Modified Caregiver Strain Index. The tool has 13 questions that measure strain related to care provision. Scoring is 2 points for each 'yes', 1 point for each 'sometimes', and 0 for each 'no' response. Scoring ranges from 26 to 0; a higher score indicates a higher level of caregiver strain.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Caregiver Stress
Description: Caregiver stress will be assessed by the Caregiver Self-Assessment Questionnaire. This questionnaire is 18 questions, 16 with yes or no responses, and 2 ranking questions. Typically a higher score indicates a higher level of caregiver stress.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Caregiver Quality of Life
Description: Caregiver quality of life will be assessed by the Adult Carer Quality of Life Questionnaire. The Adult Carer Quality of Life Questionnaire is a 40-item instrument that measures the overall quality of life for adult carers. Scores on the have a possible range of 0 to 120 with higher scores indicating greater quality of life.
Time Frame: Baseline to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: Events collected during outcome assessment appointments, before each exercise session, and during monthly health education meetings.
Arm/Group | Remote High | Remote Low | Personal Coach
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/34 | 3/32 | 1/15
Other Adverse Events (participants affected / at risk) | 7/34 | 1/32 | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remote High (N=34) | Remote Low (N=32) | Personal Coach (N=15)
Cholecystectomy (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Emergent gall bladder removal
Mitral Valve Regurgitation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Transespophageal echocardiogram revealed severe mitral valve regurgitation related to congenital heart disease
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Hospital admittance due to pulmonary edema cause by congestive heart failure
Appendectomy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — Emergent appendectomy due to ruptured appendix
Spinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Surgery to mitigate effects of spinal infection.
Isthmic Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Surgery to mitigate the effects of previous isthmus spondylolisthesis.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remote High (N=34) | Remote Low (N=32) | Personal Coach (N=15)
Ankle Injury (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2)
COVID-19 Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis and gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT04048759/Prot_SAP_000.pdf